CLINICAL TRIAL: NCT00904774
Title: Polymorphisms of Genes Controlling Alveolar Development and Risk of Bronchopulmonary Dysplasia
Brief Title: Genetic Susceptibility for Bronchopulmonary Dysplasia in Preterm Infants
Acronym: GENBPD
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Delacourt, Christophe, MD, PhD, INSERM U955
Other Study IDs: AOR 07 018
Record Dates: First submitted 2009-05-19; First posted 2009-05-20 (Estimated); Last update posted 2009-05-20 (Estimated); Status verified 2009-05

CONDITIONS: Bronchopulmonary Dysplasia
Keywords: bronchopulmonary dysplasia; neonates; lung development; prematurity
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- premature neonates: gestational age less than 28 weeks

SUMMARY:
Despite considerable obstetric and neonatal advances in the care of very low birth weight (VLBW) neonates, bronchopulmonary dysplasia (BPD) continues to occur among 20 to 40% of surviving infants, and new ways for combatting this disease must be found. BPD appears to result from arrested lung development, but its etiology has not yet been fully established. Besides the role of the exposure of the immature lung to injurious factors in the development of BPD, a genetic susceptibility for BPD in preterm infants was recently evidenced. Taking advantage of new genomic technologies, the objective of the investigators' project is to identify predisposing human genetic variants through:

1. a genome-wide association (GWA) study in VLBW neonates,
2. a candidate-gene association study, including selection of single nucleotide polymorphisms (SNPs) found in (a) and
3. functional studies of any SNP found to be convincingly associated with BPD in (a) and (b).

ELIGIBILITY:
Inclusion Criteria:

* Gestational age < 28 weeks
* Inborn birth
* Prophylactic administration of surfactant in the delivery room
* Written informed consent obtained from parents

Exclusion Criteria:

* Gestational age of 28 weeks or more
* Outborn birth
* No prophylactic administration of surfactant in the delivery room
* Congenital malformation
* Absence of written informed consent obtained from parents

Max Age: 8 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Premature neonates
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2009-05

PRIMARY OUTCOMES:
bronchopulmonary dysplasia | 36 weeks of postconceptional age

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Intercommunal, Créteil, France

REFERENCES:
- [Background] Hadchouel A, Decobert F, Franco-Montoya ML, Halphen I, Jarreau PH, Boucherat O, Martin E, Benachi A, Amselem S, Bourbon J, Danan C, Delacourt C. Matrix metalloproteinase gene polymorphisms and bronchopulmonary dysplasia: identification of MMP16 as a new player in lung development. PLoS One. 2008 Sep 11;3(9):e3188. doi: 10.1371/journal.pone.0003188. PMID 18784838
- See also: The french PremUp Foundation is dedicated to pregnancy and the newborn — http://www.premup.org/